CLINICAL TRIAL: NCT04170413
Title: Feasibility of Using CeVUS During Urodynamic Studies
Brief Title: Feasibility of Using Contrast Enhanced Voiding Urosonography (CeVUS) During Urodynamic Studies
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Reza Daugherty, MD, Associate Professor of Radiology and Pediatrics, University of Virginia
Other Study IDs: 14717
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Neurogenic Bladder
Keywords: contrast ultrasound; urodynamics
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CeVUS Urodynamic: patients undergoing urodynamic study with CeVUS
  Interventions: Drug: CeVUS

INTERVENTIONS:
Drug: CeVUS — Contrast enhanced voiding urosonography

SUMMARY:
The investigators will assess the feasibility of replacing fluoroscopy/iodinated contrast with ultrasound/sulfur hexafluoride lipid-type A microspheres during routine urodynamic studies.

DETAILED DESCRIPTION:
Urodynamic studies routinely involve instillation of iohexol (OmnipaqueTM), a low osmolality contrast agent, into the bladder followed by fluoroscopic imaging to assess for reflux or variant anatomy of the genitourinary system. Recently, sulfur hexafluoride lipid-type A microspheres (LumasonTM), an ultrasound contrast agent, has been approved in the United States for intravesicular administration in the pediatric population. Contrast enhanced voiding urosonography (CEvUS) is being increasingly utilized in the place of voiding cystourethrograms, with the major advantages being decreased (zero) radiation for the patient, as well as decreased cost. Given the similarity in procedure between urodynamic studies (UDS) and voiding cystourethrograms, the investigators hypothesize that a urodynamic study may be performed with contrast enhanced ultrasound instead of fluoroscopy. The investigators plan to conduct a small feasibility study by recruiting a group of 30 patients under the age of 18, who are willing to undergo their normally scheduled UDS in addition to CEvUS. The UDS typically consists of two cycles of bladder filling and voiding; the investigators intend to replace the use of fluoroscopy and iohexol with ultrasound and sulfur hexafluoride lipid-type A microspheres. This will decrease the time commitment and eliminate radiation exposure for the patient. There will not be a formal analysis of data as the investigators are planning to test the feasibility of the procedure rather than gather any quantitative data. The goal of the study is to eventually implement CEvUS instead of fluoroscopy in all urodynamic and voiding studies if it is found to be a reasonable alternative. This will decrease pediatric radiation exposure, which will be especially important in the patients undergoing several studies each year.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18
* Must have had prior urodynamic study at University of Virginia

Exclusion Criteria:

* Pregnant women
* Fetuses
* Neonates
* Prisoners
* Subjects with preexisting cardiac conditions (such as heart failure and ventricular arrhythmias)
* Subjects with a known hypersensitivity to Lumason

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients presenting to UVA Pediatric Urology for follow up or repeat urodynamics study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with successful completion of urodynamics | After enrollment of 30 patients, estimated 1 year
  All usual information gathered during urodynamics was able to be obtained

CONTACTS AND LOCATIONS:
Overall Officials: Reza Daugherty, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States